CLINICAL TRIAL: NCT02900313
Title: Predictive Interest of Serum Phosphorus Level in the Early Diagnosis of Acute Renal Insufficiency in Post-operative Immediate at Patients Having Benefited From a Cardiac Surgery.
Brief Title: Serum Phosphatemia Predictive Marker for AKI Diagnosis After Cardiac Surgery
Acronym: PhosphoIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UF9585; 2015-A00781-48 (Other: ID-RCB)
Record Dates: First submitted 2016-08-16; First posted 2016-09-14 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2015-06

CONDITIONS: Cardiac Surgery With Cardiopulmonary Bypass; Complete Serum Phosphorus Measure; Complete Serum Creatinine Measure
Keywords: acute kidney injury; cardiac surgery; cardiac surgery associated acute kidney injury; renal replacement therapy; renal recovery; serum hyperphosphatemia
MeSH Terms: conditions — Acute Kidney Injury | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients having cardiac surgery (Other): Cohort of patients who are more than 18 years having cardiac surgery and having benefited from a dosage of serum phosphorus level and serum creatinine during all the duration of the hospitalisation
  Interventions: Other: cardiac surgery

INTERVENTIONS:
Other: cardiac surgery — Cohort of patients who are more than 18 years having cardiac surgery and having benefited from a dosage of serum phosphorus level and serum creatinine during all the duration of the hospitalisation

SUMMARY:
Cardiac surgery associated acute kidney injury is an independent factor of morbidity and mortality . Despite its delayed elevation, serum creatinine (Cr) remains the goal standard to diagnose AKI. Hyperphosphatemia is well-know in case of AKI because of its excretion decrease. Moreover, serum phosphorus (Ph) is daily measure d after cardiac surgery since its variation may lead to cardiac dysfunction. In case of AKI, Ph may reflect the decrease of renal function in this context. Consequently, the purpose of this study is to evaluate the predictibility of Ph to detect both AKI induction and in a second time, renal recovery.

DETAILED DESCRIPTION:
It is a one-year prospective diagnostic validation study included all patients > 18 years-odl admitted in our center after cardiac surgery. AKI is define according to KDIGO criteria and classified in the groups of severity according to the Cr elevation and the need of renal replacement therapy. Serum Cr and Ph are measured at baseline before surgery , at ICU admission, every 12 hours until ICU discharge and every 24 hours until hospital discharge. To evaluate the predictability of Of Ph to diagnose AKI, the postoperative Ph percentage of maximal elevation (%EPh) will be calculated. Then the diagnostic performance of %EPh wil be assessed by calculating the areas under the Receiver Operating Characteristic Curve (AUC) to determine an optimal threshold with sensibility, specificity, positive predictive value and negative predictive value.

ELIGIBILITY:
Inclusion Criteria:

* All the patients who are more than 18 years having cardiac surgery and having benefited from a dosage of serum phosphorus level and serum creatinine during all the duration of the hospitalisation

Exclusion Criteria:

* Chronic renal insufficiency with a glomerular filtration rate = 15ml / min / 1.73m2
* Chronic Renal insufficiency dialysed
* History of single kidney or nephrectomy
* Vulnerable people according to the article L1121-6 of the public health Code
* Protected adult or in the incapacity to give his consent according to the article L1121-8 of the public health Code
* The patient present formalizes his opposition for the continuation of the study
* Pregnant or breast-feeding Women according to the article L1121-5 of the Public health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Dosage of phosphorus | 48 hour after cardiac surgery
  Kinetic phosphorus during acute renal failure in postoperative cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marine SAOUR, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Hôpital Arnaud de Villeneuve, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided